CLINICAL TRIAL: NCT02699359
Title: Indirect Intracranial Pressure Measurement in Patients With Suspected or Documented Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HeadSense Medical (Industry)
Collaborators: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-022
Record Dates: First submitted 2016-02-22; First posted 2016-03-04 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2016-12

CONDITIONS: Brain Concussion; Brain Injuries
Keywords: concussion; mild traumatic brain injuries
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): Study participants will receive HS-1000 ICP readings for a continuous 16 minute interval in a 30 degree supine position. Recordings will be obtained in one session. When possible, these recordings will be obtained at their initial examination and all follow-up visits. Sports Medicine staff will coordinate the HS-1000 device earplug insertion and recordings so as not to interfere with, nor marginally delay the patient's normal, routine clinical evaluation.
  Interventions: Device: HS-1000 recording

INTERVENTIONS:
Device: HS-1000 recording

SUMMARY:
The HS-1000 is an innovative non-invasive monitoring device that employs advanced acoustic signal analysis to calculate ICP on a continuous basis. Initial HS-1000 clinical data also shows promise in assessing a variety of cerebral hemodynamic parameters such as cerebral blood-flow, auto regulation monitoring, and cerebrovascular vessels compliance. In the absence of a non-invasive monitor of intracranial pressure (ICP), the relationships, if any, that may exist between concussion, timing of the concussion (e.g. acute, resolving, resolved) and ICP is unknown. The new HS-1000 non-invasive device may provide insight into assessment of possible ICP changes following concussion in children.

DETAILED DESCRIPTION:
Unlike fractures, concussion can be difficult to recognize and diagnose, given lack of specific diagnostic tests or clinical findings. Current diagnostic recommendations include a multi-factorial approach involving symptom inventory, baseline and post-injury neuropsychological assessment, and balance testing.

Lacking from this paradigm is a truly objective measure of physiological changes associated with concussion. In addition, post-concussion symptoms are unique to each individual and vary in occurrence, degree, and severity. For these reasons, a clinical diagnosis of concussion should be made by a healthcare provider familiar with the athlete and knowledgeable in concussion symptom recognition and evaluation.

This study aims to determine ICP measurements derived from the HS-1000 non-invasive device in children and adolescents seen in the Akron Children's Hospital Sports Medicine Clinic for concussion (anytime during their care) compared to ICP values obtained in age and gender matched Akron Children's Hospital Sports Medicine Clinic patients with no history of head injury.

Patients with a history and/or symptoms of head trauma cared for in the Akron Children's Hospital Sports Medicine Clinic will be invited to participate in this study. Study participants will receive HS-1000 ICP readings for a continuous 16 minute interval in a 30 degree supine position. Recordings will be obtained in one session. When possible, these recordings will be obtained at their initial examination and all follow-up visits. Sports Medicine staff will coordinate the HS-1000 device earplug insertion and recordings so as not to interfere with, nor marginally delay the patient's normal, routine clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All patients 12 to < 18 years of age being seen for, diagnosed with, and/or treated for traumatic brain injury (TBI) at the Akron Children's Hospital Sports Medicine Concussion Clinic are eligible for enrollment in this study.
* The control group will consist of demographically comparable patients being treated at the Akron Children's Hospital Sports Medicine Center unrelated to head trauma. These non-brain injured study participants will receive the same ICP monitoring device measurements at their initial examination and follow-up visits as performed in concussed patients.

Exclusion Criteria:

* Receiving therapy for otitis media
* Subject with bony abnormality of the skull secondary to previous fracture or other cause that may impede HeadSense device
* Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
* For females of childbearing potential: pregnancy (positive pregnancy test)
* Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
* Any condition that may jeopardize study participation or interpretation of study results (e.g., abnormal clinical finding), or may impede the ability to obtain informed consent (e.g., developmental delay of patient or caretaker)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of recordings that correlate to concussion diagnosis using current standards | 16 minute recording period

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Congeni, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No